CLINICAL TRIAL: NCT02124161
Title: A Phase 4, Randomized, Double-blind Trial To Evaluate The Immunogenicity And Safety Of A 13-valent Pneumococcal Conjugate Vaccine When Administered Concomitantly With Seasonal Inactivated Influenza Vaccine In Adults 50 Years And Older Who Received 1 Or More Doses Of 23-valent Pneumococcal Polysaccharide Vaccine Prior To Study Enrollment.
Brief Title: Concomitant Administration of 13-valent Pneumococcal Conjugate Vaccine (13vPnC) With Influenza Vaccine in 23-valent Pneumococcal Polysaccharide (23vPS) Pre-vaccinated Adults.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Masking: Triple | Purpose: Basic Science
Other Study IDs: B1851138
Record Dates: First submitted 2014-04-24; First posted 2014-04-28 (Estimated); Results first posted 2016-07-01 (Estimated); Last update posted 2016-07-01 (Estimated); Status verified 2016-04

CONDITIONS: PREVENTION OF INVASIVE PNEUMOCOCCAL DISEASE
Keywords: Pneumococcal polysaccharide vaccine; 13-valent pneumococcal conjugate vaccine; invasive pneumococcal disease; flu vaccine
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 13vPnC+SIIV/Placebo (Other)
  Interventions: Biological: 13-valent pneumococcal conjugate vaccine; Biological: Seasonal Inactivated Influenza Vaccine; Other: Placebo
- Placebo+SIIV/13vPnC (Other)
  Interventions: Other: Placebo; Biological: Seasonal Inactivated Influenza Vaccine; Biological: 13-valent pneumococcal conjugate vaccine

INTERVENTIONS:
Biological: 13-valent pneumococcal conjugate vaccine — One (1) dose (0.5 mL) will be administered intramuscularly into the left deltoid either at Visit 1 or at Visit 2, depending on the randomization group assigned to the subject.
  Other Names: 13vPnC
  Arms: 13vPnC+SIIV/Placebo
Biological: Seasonal Inactivated Influenza Vaccine — One (1) dose of SIIV will be administered intramuscularly into the right deltoid of all subjects at Visit 1.
  Other Names: SIIV
  Arms: 13vPnC+SIIV/Placebo
Other: Placebo — One (1) dose (0.5 mL) will be administered intramuscularly into the left deltoid either at Visit 1 or at Visit 2, depending on the randomization group assigned to the subject.
  Arms: 13vPnC+SIIV/Placebo
Other: Placebo — One (1) dose (0.5 mL) will be administered intramuscularly into the left deltoid either at Visit 1 or at Visit 2, depending on the randomization group assigned to the subject.
  Arms: Placebo+SIIV/13vPnC
Biological: Seasonal Inactivated Influenza Vaccine — One (1) dose of SIIV will be administered intramuscularly into the right deltoid of all subjects at Visit 1.
  Other Names: SIIV
  Arms: Placebo+SIIV/13vPnC
Biological: 13-valent pneumococcal conjugate vaccine — One (1) dose (0.5 mL) will be administered intramuscularly into the left deltoid either at Visit 1 or at Visit 2, depending on the randomization group assigned to the subject.
  Other Names: 13vPnC
  Arms: Placebo+SIIV/13vPnC

SUMMARY:
The purpose of this study is to evaluate the immunogenicity and safety of 13-valent pneumococcal polysaccharide vaccine when given concomitantly with seasonal inactivated influenza vaccine to adults 50 years and older who have previously received 23-valent pneumococcal polysaccharide vaccine.

ELIGIBILITY:
Inclusion Criteria:

1. Evidence of a personally signed and dated informed consent document (ICD) indicating that the subject has been informed of all pertinent aspects of the study.
2. Male or female adults 50 years of age or older.
3. Documented vaccination with 1 or more prior doses of 23vPS, the last given at least 1 year prior to study enrollment.
4. Negative urine pregnancy test for all female subjects who are of child bearing potential.

Exclusion Criteria:

1. Previous vaccination with Prevnar®, Prevnar 13®, or any other investigational pneumococcal conjugate vaccine.
2. History of severe adverse reactions associated with any vaccine or vaccine-related component.
3. Allergic to egg proteins (egg or egg products) and chicken proteins.
4. History of Guillain-Barré syndrome.
5. Vaccination with any influenza vaccine within 6 months (182 days) before investigational product administration.
6. Documented S pneumoniae infection within the past 5 years before investigational product administration.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 882 (Actual)
Dates: Start 2014-09; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (44):
- United States (44):
  - Achieve Clinical Research, LLC, Birmingham, Alabama
  - Optimal Research (Formerly Accelovance), Huntsville, Alabama
  - Radiant Research, Inc., Scottsdale, Arizona
  - Kaiser Permanente Vaccine Study Center, Oakland, California
  - Kaiser Permanante South. Sacramento, Sacramento, California
  - Benchmark Research, San Francisco, California
  - Kaiser Pemanente Santa Clara, Santa Clara, California
  - Avail Clinical Research, LLC, DeLand, Florida
  - Westside Center for Clinical Research, Jacksonville, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Radiant Research, Inc., Pinellas Park, Florida
  - Meridian Clinical Research, Savannah, Georgia
  - Optimal Research, LLC, Mishawaka, Indiana
  - Clinical Research Advantage, Inc/Ridge Family Practice, Council Bluffs, Iowa
  - Johnson County Clin-Trials, Inc., Lenexa, Kansas
  - Benchmark Research, Metairie, Louisiana
  - Meridian Clinical Research, Bellevue, Nebraska
  - Meridian Clinical Research, Norfolk, Nebraska
  - Meridian Clinical Research, LLC, Omaha, Nebraska
  - Clinical Research Center of Nevada, LLC, Las Vegas, Nevada
  - Clinical Research Advantage, Inc., Las Vegas, Nevada
  - United Medical Associates, Binghamton, New York
  - Regional Clinical Research, Inc., Endwell, New York
  - Rochester Clinical Research, Inc., Rochester, New York
  - PMG Research of Raleigh, LLC d/b/a PMG Research of Cary, Cary, North Carolina
  - PharmQuest, Greensboro, North Carolina
  - PMG Research of Hickory, LLC, Hickory, North Carolina
  - Clinical Trials of America, Inc., Winston-Salem, North Carolina
  - PMG Research of Winston-Salem, Winston-Salem, North Carolina
  - Radiant Research, Inc, Columbus, Ohio
  - Prestige Clinical Research, Franklin, Ohio
  - Preferred Primary Care Physicians, Inc., Carnegie, Pennsylvania
  - Brandywine Clinical Research, Downingtown, Pennsylvania
  - Omega Medical Research, Warwick, Rhode Island
  - PMG Research of Charleston, Mt. Pleasant, South Carolina
  - Internal Medicine and Pediatric Associates of Bristol, PC, Bristol, Tennessee
  - Volunteer Research Group, Knoxville, Tennessee
  - Benchmark Research, Austin, Texas
  - Benchmark Research, Fort Worth, Texas
  - Diagnostics Research Group, San Antonio, Texas
  - Radiant Research, Inc., Murray, Utah
  - J. Lewis Research, Inc. / Foothill Family Clinic, Salt Lake City, Utah
  - J. Lewis Research, Inc. / Foothill Family Clinic South, Salt Lake City, Utah
  - J. Lewis Research, Inc. / Jordan River Family Medicine, South Jordan, Utah

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1851138&StudyName=Concomitant%20administration%20of%2013-valent%20Pneumococcal%20Conjugate%20Vaccine%20%2813vPnC%29%20with%20influenza%20vaccine%20in%2023-valent%20Pneumococcal%20Polysaccharid

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 882 participants who were greater than or equal to (>=) 50 years of age and previously vaccinated with at least 1 dose of 23-valent pneumococcal polysaccharide vaccine (23vPS) were randomized in this study but 6 participants (2 participants in 13vPnC+QIV/Placebo arm and 4 participants in Placebo+QIV/13vPnC arm) were randomized but not vaccinated.
Groups:
- 13vPnC+QIV/Placebo: Participants received 0.5 milliliter (mL) single dose of 13-valent pneumococcal conjugate (13vPnC) vaccine intramuscularly along with a dose of quadrivalent influenza vaccine (QIV, as per official recommendations) intramuscularly at Day 1 (Vaccination 1) followed by 0.5 mL placebo matched to 13vPnC vaccine intramuscularly 1 month after Vaccination 1.
- Placebo+QIV/13vPnC: Participants received 0.5 mL placebo matched to 13vPnC vaccine intramuscularly along with a dose of QIV intramuscular injection as per official recommendations at Day 1 (Vaccination 1) followed by 0.5 mL single dose of 13vPnC vaccine intramuscularly 1 month after Vaccination 1.
Period: Overall Study
Arm/Group | 13vPnC+QIV/Placebo | Placebo+QIV/13vPnC
Started | 441 | 441
Vaccination 1 | 439 | 437
Vaccination 2 | 431 | 432
Completed | 425 | 426
Not Completed | 16 | 15
Not completed — Other unspecified | 0 | 1
Not completed — Death | 1 | 0
Not completed — Protocol Violation | 2 | 1
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Adverse Event | 2 | 0
Not completed — Does not meet entrance criteria | 2 | 3
Not completed — No longer meets eligibility criteria | 5 | 4
Not completed — Lost to Follow-up | 3 | 4

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who received at least 1 dose of vaccination.
Groups:
- Total: Total of all reporting groups
Arm/Group | 13vPnC+QIV/Placebo | Placebo+QIV/13vPnC | Total
Number analyzed (Participants) | 439 | 437 | 876
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.9 (9) | 66.4 (8.85) | 66.7 (8.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 234 | 249 | 483
  Male | 205 | 188 | 393

OUTCOME MEASURES:

1. Primary Outcome: Serotype-specific Opsonophagocytic Activity (OPA) Geometric Mean Titers (GMTs) for 13 Pneumococcal Serotypes
Description: Serotype-specific OPA GMTs for each of the 13 pneumococcal common serotypes (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F) were logarithmically transformed for analysis. Confidence intervals (CIs) for GMT were back-transformed based on the Student t distribution for the mean logarithm of the titers. GMTs were calculated using all participants with available data for the specified blood draw. Here, "number of participants analyzed" signifies the participants who were evaluable at this timepoint and "n" signifies participants with a determinate OPA titer to the given serotype.
Time Frame: 1 month after Vaccination 1 for 13vPnC+QIV/Placebo, 1 Month After Vaccination 2 for Placebo+QIV/13vPnC
Population: Evaluable immunogenicity population: eligible, randomized participants of 50 years of age or above, received all study vaccinations in assigned sequence with expected concomitant vaccination, had at least 1 valid, determinate assay results, had pre and post vaccination blood drawn within protocol-specified time frames, no major protocol violations.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | 13vPnC+QIV/Placebo | Placebo+QIV/13vPnC
Number analyzed (Participants) | 427 | 425
titer
  Serotype 1 (n= 419, 417) | 75 [65.0 to 87.0] | 83 [71.1 to 96.1]
  Serotype 3 (n= 422, 418) | 41 [36.2 to 46] | 49 [43.6 to 55.3]
  Serotype 4 (n= 412, 417) | 587 [489.9 to 702.5] | 824 [692.2 to 980]
  Serotype 5 (n= 423, 414) | 97 [83.8 to 111.7] | 101 [86.6 to 117.2]
  Serotype 6A (n= 420, 415) | 953 [805.7 to 1126.3] | 1413 [1203.3 to 1659.4]
  Serotype 6B (n= 414, 405) | 867 [722.3 to 1039.6] | 1041 [860.5 to 1260]
  Serotype 7F (n= 424, 419) | 651 [582.4 to 728] | 670 [599.7 to 748.5]
  Serotype 9V (n= 419, 415) | 699 [613.7 to 797.2] | 838 [734.2 to 957.5]
  Serotype 14 (n= 421, 416) | 574 [496.8 to 663] | 760 [665.6 to 868]
  Serotype 18C (n= 420, 414) | 713 [598.9 to 849.9] | 865 [726.4 to 1030.5]
  Serotype 19A (n= 425, 419) | 337 [294.9 to 384.6] | 390 [344.4 to 441.1]
  Serotype 19F (n= 423, 416) | 324 [274.8 to 382.5] | 360 [302.7 to 427.9]
  Serotype 23F (n= 421, 417) | 278 [223.9 to 344.7] | 364 [294.3 to 451.3]
Statistical Analysis 1: Comparison: 13vPnC+QIV/Placebo vs Placebo+QIV/13vPnC; Serotype 1: Confidence Intervals (CIs) for the ratio were back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC+QIV/placebo - placebo+QIV/13vPnC); Test type: Non-Inferiority or Equivalence — The criterion for noninferiority was the lower bound of the 2-sided 95% CI for the GMT ratio was greater than 0.5 (2-fold criterion); GMT Ratio = 0.9, 95% CI 2-sided [0.74 to 1.12]
Statistical Analysis 2: Comparison: 13vPnC+QIV/Placebo vs Placebo+QIV/13vPnC; Serotype 3: Confidence Intervals (CIs) for the ratio were back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC+QIV/placebo - placebo+QIV/13vPnC); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; GMT Ratio = 0.8, 95% CI 2-sided [0.70 to 0.98]
Statistical Analysis 3: Comparison: 13vPnC+QIV/Placebo vs Placebo+QIV/13vPnC; Serotype 4: Confidence Intervals (CIs) for the ratio were back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC+QIV/placebo - placebo+QIV/13vPnC); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; GMT Ratio = 0.7, 95% CI 2-sided [0.55 to 0.91]
Statistical Analysis 4: Comparison: 13vPnC+QIV/Placebo vs Placebo+QIV/13vPnC; Serotype 5: Confidence Intervals (CIs) for the ratio were back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC+QIV/placebo - placebo+QIV/13vPnC); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; GMT Ratio = 1.0, 95% CI 2-sided [0.78 to 1.18]
Statistical Analysis 5: Comparison: 13vPnC+QIV/Placebo vs Placebo+QIV/13vPnC; Serotype 6A: Confidence Intervals (CIs) for the ratio were back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC+QIV/placebo - placebo+QIV/13vPnC); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; GMT Ratio = 0.7, 95% CI 2-sided [0.53 to 0.85]
Statistical Analysis 6: Comparison: 13vPnC+QIV/Placebo vs Placebo+QIV/13vPnC; Serotype 6B: Confidence Intervals (CIs) for the ratio were back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC+QIV/placebo - placebo+QIV/13vPnC); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; GMT Ratio = 0.8, 95% CI 2-sided [0.64 to 1.08]
Statistical Analysis 7: Comparison: 13vPnC+QIV/Placebo vs Placebo+QIV/13vPnC; Serotype 7F: Confidence Intervals (CIs) for the ratio were back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC+QIV/placebo - placebo+QIV/13vPnC); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; GMT Ratio = 1.0, 95% CI 2-sided [0.83 to 1.14]
Statistical Analysis 8: Comparison: 13vPnC+QIV/Placebo vs Placebo+QIV/13vPnC; Serotype 9V: Confidence Intervals (CIs) for the ratio were back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC+QIV/placebo - placebo+QIV/13vPnC); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; GMT Ratio = 0.8, 95% CI 2-sided [0.69 to 1.0]
Statistical Analysis 9: Comparison: 13vPnC+QIV/Placebo vs Placebo+QIV/13vPnC; Serotype 14: Confidence Intervals (CIs) for the ratio were back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC+QIV/placebo - placebo+QIV/13vPnC); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; GMT Ratio = 0.8, 95% CI 2-sided [0.62 to 0.92]
Statistical Analysis 10: Comparison: 13vPnC+QIV/Placebo vs Placebo+QIV/13vPnC; Serotype 18C: Confidence Intervals (CIs) for the ratio were back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC+QIV/placebo - placebo+QIV/13vPnC); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; GMT Ratio = 0.8, 95% CI 2-sided [0.64 to 1.06]
Statistical Analysis 11: Comparison: 13vPnC+QIV/Placebo vs Placebo+QIV/13vPnC; Serotype 19A: Confidence Intervals (CIs) for the ratio were back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC+QIV/placebo - placebo+QIV/13vPnC); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; GMT Ratio = 0.9, 95% CI 2-sided [0.72 to 1.04]
Statistical Analysis 12: Comparison: 13vPnC+QIV/Placebo vs Placebo+QIV/13vPnC; Serotype 19F: Confidence Intervals (CIs) for the ratio were back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC+QIV/placebo - placebo+QIV/13vPnC); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; GMT Ratio = 0.9, 95% CI 2-sided [0.71 to 1.14]
Statistical Analysis 13: Comparison: 13vPnC+QIV/Placebo vs Placebo+QIV/13vPnC; Serotype 23F: Confidence Intervals (CIs) for the ratio were back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC+QIV/placebo - placebo+QIV/13vPnC); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; GMT Ratio = 0.8, 95% CI 2-sided [0.56 to 1.03]

2. Primary Outcome: Hemagglutination Inhibition Assay (HAI) Geometric Mean Titers (GMTs) for Each Influenza Virus Strain in Quadrivalent Influenza Vaccine (QIV)
Description: HAI GMTs were computed for assay titers collected 1 month after Vaccination 1 by vaccine sequence for each influenza virus strain (A/H1N1, A/H3N2, B/Brisbane and B/Massachusetts). CIs were back-transformations of a CI based on the Student t distribution for the mean logarithm of the titers. HAI GMTs were calculated using all participants with available data for the specified blood draw. Here, "number of participants analyzed" signifies participants with a determinate HAI titer to the given strain.
Time Frame: 1 month after Vaccination 1
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | 13vPnC+QIV/Placebo | Placebo+QIV/13vPnC
Number analyzed (Participants) | 427 | 430
titer
  Strain: A/H1N1 | 115 [104.0 to 126.8] | 113 [101.6 to 124.7]
  Strain: A/H3N2 | 226 [206.1 to 248.5] | 196 [178.0 to 216.1]
  Strain: B/Brisbane | 28 [25.7 to 31.0] | 26 [23.7 to 28.7]
  Strain: B/Massachusetts | 45 [41.0 to 50.3] | 43 [39.1 to 48.2]
Statistical Analysis 1: Comparison: 13vPnC+QIV/Placebo vs Placebo+QIV/13vPnC; Strain A/H1N1: CIs for the ratio were back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC+QIV/placebo - placebo+QIV/13vPnC); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; GMT Ratio = 1.0, 95% CI 2-sided [0.88 to 1.18]
Statistical Analysis 2: Comparison: 13vPnC+QIV/Placebo vs Placebo+QIV/13vPnC; Strain A/H3N2: CIs for the ratio were back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC+QIV/placebo - placebo+QIV/13vPnC); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; GMT Ratio = 1.2, 95% CI 2-sided [1.01 to 1.32]
Statistical Analysis 3: Comparison: 13vPnC+QIV/Placebo vs Placebo+QIV/13vPnC; Strain B/Brisbane: CIs for the ratio were back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC+QIV/placebo - placebo+QIV/13vPnC); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; GMT Ratio = 1.1, 95% CI 2-sided [0.95 to 1.24]
Statistical Analysis 4: Comparison: 13vPnC+QIV/Placebo vs Placebo+QIV/13vPnC; Strain B/Massachusetts: CIs for the ratio were back transformations of CI based on the Student t distribution for the mean difference of the logarithms of the measures (13vPnC+QIV/placebo - placebo+QIV/13vPnC); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; GMT Ratio = 1.0, 95% CI 2-sided [0.90 to 1.21]

3. Primary Outcome: Percentage of Participants With Treatment--Emergent Adverse Events (AEs) or Serious Adverse Events (SAEs) After Vaccination 1
Description: An AE was any untoward medical occurrence in a participant who received vaccine without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. AEs included both SAEs and non-serious adverse events (Non-SAEs).
Time Frame: Within 28 to 42 days after Vaccination 1
Population: Safety population included all participants who received at least 1 dose of vaccination.
Measure: Number; unit: percentage of participants
Arm/Group | 13vPnC+QIV/Placebo | Placebo+QIV/13vPnC
Number analyzed (Participants) | 439 | 437
percentage of participants
  AE | 15.3 | 11.9
  SAE | 1.4 | 0

4. Primary Outcome: Percentage of Participants With Treatment--Emergent Adverse Events (AEs) or Serious Adverse Events (SAEs) After Vaccination 2
Description: as for outcome 3
Time Frame: Within 28 to 42 days after Vaccination 2
Population: Safety population included all participants who received at least 1 dose of vaccination. Here, "number of participants analyzed" signifies participants who were evaluable at this timepoint.
Measure: Number; unit: percentage of participants
Arm/Group | 13vPnC+QIV/Placebo | Placebo+QIV/13vPnC
Number analyzed (Participants) | 431 | 432
percentage of participants
  AE | 10.4 | 12.5
  SAE | 1.6 | 1.4

5. Primary Outcome: Percentage of Participants With Treatment--Emergent Adverse Events (AEs) or Serious Adverse Events (SAEs) After 13vPnC Vaccination
Description: as for outcome 3
Time Frame: Baseline (Vaccination 1) up to 28 to 42 Days after Vaccination 2
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | 13vPnC+QIV/Placebo | Placebo+QIV/13vPnC
Number analyzed (Participants) | 439 | 432
percentage of participants
  AE | 15.3 | 12.5
  SAE | 1.4 | 1.4
Statistical Analysis 1: Comparison: 13vPnC+QIV/Placebo vs Placebo+QIV/13vPnC; AE: Exact 2-sided confidence interval (based on Chan and Zhang) for the difference in proportions, 13vPnC+QIV /placebo - placebo+QIV/13vPnC, expressed as a percentage; Test type: Superiority or Other; Percentage Difference = 2.8, 95% CI 2-sided [-1.9 to 7.4]
Statistical Analysis 2: Comparison: 13vPnC+QIV/Placebo vs Placebo+QIV/13vPnC; SAE: Exact 2-sided confidence interval (based on Chan and Zhang) for the difference in proportions, 13vPnC+QIV /placebo - placebo+QIV/13vPnC, expressed as a percentage; Test type: Superiority or Other; Percentage Difference = -0.0, 95% CI 2-sided [-1.8 to 1.7]

6. Primary Outcome: Percentage of Participants With Treatment--Emergent Adverse Events (AEs) or Serious Adverse Events (SAEs) at the 6-Month Follow-up
Description: as for outcome 3
Time Frame: Within 168 to 196 days after Vaccination 2
Population: Safety population included all participants who received at least 1 dose of vaccination.
Measure: Number; unit: percentage of participants
Arm/Group | 13vPnC+QIV/Placebo | Placebo+QIV/13vPnC
Number analyzed (Participants) | 439 | 437
percentage of participants
  AE | 2.5 | 2.7
  SAE | 1.1 | 1.4

7. Secondary Outcome: Percentage of Participants Achieving Pneumococcal Serotype-specific Opsonophagocytic Activity (OPA) Antibody Titer Greater Than or Equal to (>=) Lower Limit of Quantitation (LLOQ)
Description: Percentage of participants achieving predefined OPA antibody titer >= LLOQ for each of the 13 pneumococcal serotypes (LLOQs for each serotype OPA were set as- serotype 1: 18; serotype 3: 12; serotype 4: 21; serotype 5: 29; serotype 6A: 37; serotype 6B: 43; serotype 7F: 210; serotype 9V: 345; serotype 14: 35; serotype 18C: 31; serotype 19A: 18; serotype 19F: 48; and serotype 23F: 13) determined in blood samples of all participants were calculated. Exact, 2-sided 95% CIs based on the observed percentage of participants were determined by using Clopper and Pearson method. OPA titers were calculated using all participants with available data from 1 month after 13vPnC vaccination blood draw. Here, "number of participants analyzed" signifies the participants who were evaluable at this timepoint and "n" signifies participants with valid and determinate assay results to the specified serotype.
Time Frame: 1 Month After Vaccination 1 for 13vPnC+QIV/Placebo, 1 month after Vaccination 2 for Placebo+QIV/13vPnC
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 13vPnC+QIV/Placebo | Placebo+QIV/13vPnC
Number analyzed (Participants) | 427 | 425
percentage of participants
  Serotype 1 (n= 419, 417) | 77.3 [73.0 to 81.3] | 80.1 [75.9 to 83.8]
  Serotype 3 (n= 422, 418) | 79.4 [75.2 to 83.1] | 83.7 [79.8 to 87.1]
  Serotype 4 (n= 412, 417) | 88.6 [85.1 to 91.5] | 92.1 [89.1 to 94.5]
  Serotype 5 (n= 423, 414) | 74.5 [70.0 to 78.6] | 72.7 [68.1 to 76.9]
  Serotype 6A (n= 420, 415) | 90.5 [87.3 to 93.1] | 94.2 [91.5 to 96.3]
  Serotype 6B (n= 414, 405) | 85.0 [81.2 to 88.3] | 86.4 [82.7 to 89.6]
  Serotype 7F (n= 424, 419) | 82.3 [78.3 to 85.8] | 83.5 [79.6 to 87.0]
  Serotype 9V (n= 419, 415) | 65.2 [60.4 to 69.7] | 71.3 [66.7 to 75.6]
  Serotype 14 (n= 421, 416) | 91.4 [88.4 to 93.9] | 95.2 [92.7 to 97.0]
  Serotype 18C (n= 420, 414) | 88.8 [85.4 to 91.7] | 91.3 [88.2 to 93.8]
  Serotype 19A (n= 425, 419) | 95.5 [93.1 to 97.3] | 97.4 [95.4 to 98.7]
  Serotype 19F (n= 423, 416) | 79.9 [75.8 to 83.6] | 79.6 [75.4 to 83.3]
  Serotype 23F (n= 421, 417) | 80.3 [76.2 to 84.0] | 84.2 [80.3 to 87.5]
Statistical Analysis 1: Comparison: 13vPnC+QIV/Placebo vs Placebo+QIV/13vPnC; Serotype 1: Exact 2-sided CI and corresponding p-value (based on Chan and Zhang) for the difference in proportions, (13vPnC+QIV/placebo - placebo+QIV/13vPnC), expressed as a percentage; Test type: Superiority or Other; p = 0.333, Chan and Zhang method; Percentage Difference = -2.8, 95% CI 2-sided [-8.3 to 2.8]
Statistical Analysis 2: Comparison: 13vPnC+QIV/Placebo vs Placebo+QIV/13vPnC; Serotype 3: Exact 2-sided CI and corresponding p-value (based on Chan and Zhang) for the difference in proportions, (13vPnC+QIV/placebo - placebo+QIV/13vPnC), expressed as a percentage; Test type: Superiority or Other; p = 0.105, Chan and Zhang method; Percentage Difference = -4.3, 95% CI 2-sided [-9.6 to 0.9]
Statistical Analysis 3: Comparison: 13vPnC+QIV/Placebo vs Placebo+QIV/13vPnC; Serotype 4: Exact 2-sided CI and corresponding p-value (based on Chan and Zhang) for the difference in proportions, (13vPnC+QIV/placebo - placebo+QIV/13vPnC), expressed as a percentage; Test type: Superiority or Other; p = 0.090, Chan and Zhang method; Percentage Difference = -3.5, 95% CI 2-sided [-7.6 to 0.6]
Statistical Analysis 4: Comparison: 13vPnC+QIV/Placebo vs Placebo+QIV/13vPnC; Serotype 5: Exact 2-sided CI and corresponding p-value (based on Chan and Zhang) for the difference in proportions, (13vPnC+QIV/placebo - placebo+QIV/13vPnC), expressed as a percentage; Test type: Superiority or Other; p = 0.590, Chan and Zhang method; Percentage Difference = 1.8, 95% CI 2-sided [-4.2 to 7.8]
Statistical Analysis 5: Comparison: 13vPnC+QIV/Placebo vs Placebo+QIV/13vPnC; Serotype 6A: Exact 2-sided CI and corresponding p-value (based on Chan and Zhang) for the difference in proportions, (13vPnC+QIV/placebo - placebo+QIV/13vPnC), expressed as a percentage; Test type: Superiority or Other; p = 0.044, Chan and Zhang method; Percentage Difference = -3.7, 95% CI 2-sided [-7.5 to -0.1]
Statistical Analysis 6: Comparison: 13vPnC+QIV/Placebo vs Placebo+QIV/13vPnC; Serotype 6B: Exact 2-sided CI and corresponding p-value (based on Chan and Zhang) for the difference in proportions, (13vPnC+QIV/placebo - placebo+QIV/13vPnC), expressed as a percentage; Test type: Superiority or Other; p = 0.574, Chan and Zhang method; Percentage Difference = -1.4, 95% CI 2-sided [-6.2 to 3.4]
Statistical Analysis 7: Comparison: 13vPnC+QIV/Placebo vs Placebo+QIV/13vPnC; Serotype 7F: Exact 2-sided CI and corresponding p-value (based on Chan and Zhang) for the difference in proportions, (13vPnC+QIV/placebo - placebo+QIV/13vPnC), expressed as a percentage; Test type: Superiority or Other; p = 0.648, Chan and Zhang method; Percentage Difference = -1.2, 95% CI 2-sided [-6.3 to 3.9]
Statistical Analysis 8: Comparison: 13vPnC+QIV/Placebo vs Placebo+QIV/13vPnC; Serotype 9V: Exact 2-sided CI and corresponding p-value (based on Chan and Zhang) for the difference in proportions, (13vPnC+QIV/placebo - placebo+QIV/13vPnC), expressed as a percentage; Test type: Superiority or Other; p = 0.057, Chan and Zhang method; Percentage Difference = -6.2, 95% CI 2-sided [-12.5 to 0.2]
Statistical Analysis 9: Comparison: 13vPnC+QIV/Placebo vs Placebo+QIV/13vPnC; Serotype 14: Exact 2-sided CI and corresponding p-value (based on Chan and Zhang) for the difference in proportions, (13vPnC+QIV/placebo - placebo+QIV/13vPnC), expressed as a percentage; Test type: Superiority or Other; p = 0.030, Chan and Zhang method; Percentage Difference = -3.7, 95% CI 2-sided [-7.3 to -0.3]
Statistical Analysis 10: Comparison: 13vPnC+QIV/Placebo vs Placebo+QIV/13vPnC; Serotype 18C: Exact 2-sided CI and corresponding p-value (based on Chan and Zhang) for the difference in proportions, (13vPnC+QIV/placebo - placebo+QIV/13vPnC), expressed as a percentage; Test type: Superiority or Other; p = 0.233, Chan and Zhang method; Percentage Difference = -2.5, 95% CI 2-sided [-6.6 to 1.6]
Statistical Analysis 11: Comparison: 13vPnC+QIV/Placebo vs Placebo+QIV/13vPnC; Serotype 19A: Exact 2-sided CI and corresponding p-value (based on Chan and Zhang) for the difference in proportions, (13vPnC+QIV/placebo - placebo+QIV/13vPnC), expressed as a percentage; Test type: Superiority or Other; p = 0.152, Chan and Zhang method; Percentage Difference = -1.8, 95% CI 2-sided [-4.5 to 0.7]
Statistical Analysis 12: Comparison: 13vPnC+QIV/Placebo vs Placebo+QIV/13vPnC; Serotype 19F: Exact 2-sided CI and corresponding p-value (based on Chan and Zhang) for the difference in proportions, (13vPnC+QIV/placebo - placebo+QIV/13vPnC), expressed as a percentage; Test type: Superiority or Other; p = 0.926, Chan and Zhang method; Percentage Difference = 0.3, 95% CI 2-sided [-5.1 to 5.8]
Statistical Analysis 13: Comparison: 13vPnC+QIV/Placebo vs Placebo+QIV/13vPnC; Serotype 23F: Exact 2-sided CI and corresponding p-value (based on Chan and Zhang) for the difference in proportions, (13vPnC+QIV/placebo - placebo+QIV/13vPnC), expressed as a percentage; Test type: Superiority or Other; p = 0.143, Chan and Zhang method; Percentage Difference = -3.9, 95% CI 2-sided [-9.1 to 1.3]

8. Secondary Outcome: Geometric Mean Fold Rise (GMFR) for Pneumococcal Serotype-Specific Opsonophagocytic Activity (OPA) Titers 1 Month After 13vPnC Vaccination 1 to Immediately Before 13vPnC Vaccination 1
Description: GMFR for the 13 pneumococcal serotypes (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F) 1 month after Vaccination 1 to before Vaccination 1 were computed using the logarithmically transformed assay results. CIs for GMFR were back transformations of a CI based on the Student t distribution for the mean logarithm of the mean fold rise. GMFRs were calculated using all participants with available data from both before Vaccination 1 and 1 month after Vaccination 1 blood draws. Here, "n" signifies participants with valid and determinate assay results for specified serotype at both the given visits. Number of participants who received at least 1 dose of 13vPnC during Vaccination 1 were analyzed.
Time Frame: Immediately before Vaccination 1, 1 month after Vaccination 1
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: fold rise
Arm/Group | 13vPnC+QIV/Placebo
Number analyzed (Participants) | 427
fold rise
  Serotype 1 (n= 417) | 3.6 [3.20 to 4.14]
  Serotype 3 (n= 419) | 3.4 [3.05 to 3.85]
  Serotype 4 (n= 399) | 9.1 [7.33 to 11.18]
  Serotype 5 (n= 422) | 3.0 [2.70 to 3.43]
  Serotype 6A (n= 408) | 13.7 [11.30 to 16.62]
  Serotype 6B (n= 391) | 8.9 [7.29 to 10.87]
  Serotype 7F (n= 417) | 2.7 [2.40 to 2.98]
  Serotype 9V (n= 405) | 2.1 [1.92 to 2.38]
  Serotype 14 (n= 411) | 2.0 [1.78 to 2.30]
  Serotype 18C (n= 417) | 4.0 [3.38 to 4.74]
  Serotype 19A (n= 424) | 3.7 [3.20 to 4.28]
  Serotype 19F (n= 419) | 4.2 [3.60 to 4.87]
  Serotype 23F (n= 418) | 8.7 [7.07 to 10.61]

9. Secondary Outcome: Geometric Mean Fold Rise (GMFR) for Pneumococcal Serotype-Specific Opsonophagocytic Activity (OPA) Titers 1 Month After 13vPnC Vaccination 2 to Immediately Before 13vPnC Vaccination 2
Description: GMFR for the 13 pneumococcal serotypes (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F) 1 month after Vaccination 2 to before Vaccination 2 (1 month after Vaccination 1) were computed using the logarithmically transformed assay results. CIs for GMFR were back transformations of a CI based on the Student t distribution for the mean logarithm of the mean fold rise. GMFRs were calculated using all participants with available data from both before Vaccination 2 and 1 month after Vaccination 2 blood draws. Here, "number of participants analyzed" signifies total participants who were evaluable at this timepoint and "n" signifies participants with valid and determinate assay results for specified serotype at both the given visits. Number of participants who received at least 1 dose of 13vPnC during Vaccination 2 were analyzed.
Time Frame: Immediately before Vaccination 2, 1 month after Vaccination 2
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: fold rise
Arm/Group | Placebo+QIV/13vPnC
Number analyzed (Participants) | 425
fold rise
  Serotype 1 (n =413) | 3.6 [3.19 to 4.16]
  Serotype 3 (n= 414) | 3.9 [3.47 to 4.42]
  Serotype 4 (n= 391) | 10.4 [8.28 to 12.94]
  Serotype 5 (n= 411) | 3.3 [2.87 to 3.72]
  Serotype 6A (n= 399) | 17.9 [14.73 to 21.86]
  Serotype 6B (n= 382) | 9.5 [7.69 to 11.67]
  Serotype 7F (n= 407) | 2.7 [2.41 to 3.03]
  Serotype 9V (n= 399) | 2.4 [2.12 to 2.71]
  Serotype 14 (n= 406) | 2.3 [1.98 to 2.60]
  Serotype 18C (n= 408) | 6.3 [5.21 to 7.51]
  Serotype 19A (n= 416) | 4.6 [4.02 to 5.35]
  Serotype 19F (n= 410) | 4.8 [4.12 to 5.69]
  Serotype 23F (n= 412) | 12.9 [10.42 to 15.88]

10. Secondary Outcome: Percentage of Participants Achieving Seroconversion in Hemagglutination Inhibition Assay (HAI) Titers
Description: Percentage of participants achieving seroconversion in HAI titers was defined as the percentage of participants with either before Vaccination 1 (pre-vaccination 1) HAI titer less than <1:10 and after Vaccination 1 (post-vaccination 1) HAI titer >=1:40 or before Vaccination 1 (pre-vaccination 1) HAI titer >=1:10 and a minimum 4-fold rise in after Vaccination 1 (post-vaccination 1) HAI antibody titer with respect to before Vaccination 1 (pre-vaccination) titer for influenza virus strains. Here, "number of participants analyzed" signifies the participants who were evaluable at this timepoint.
Time Frame: Immediately before Vaccination 1, 1 month after Vaccination 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 13vPnC+QIV/Placebo | Placebo+QIV/13vPnC
Number analyzed (Participants) | 427 | 430
percentage of participants
  Strain: A/H1N1 | 29.3 [25.0 to 33.8] | 24.2 [20.2 to 28.5]
  Strain: A/H3N2 | 27.9 [23.7 to 32.4] | 31.6 [27.3 to 36.3]
  Strain: B/Brisbane | 21.3 [17.5 to 25.5] | 22.3 [18.5 to 26.6]
  Strain: B/Massachusetts | 23.2 [19.3 to 27.5] | 24.7 [20.6 to 29.0]
Statistical Analysis 1: Comparison: 13vPnC+QIV/Placebo vs Placebo+QIV/13vPnC; Strain A/H1N1: Exact 2-sided CI and corresponding p-value (based on Chan and Zhang) for the difference in proportions, (13vPnC+QIV/placebo - placebo+QIV/13vPnC), expressed as a percentage; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.094, Chan and Zhang method; Percentage Difference = 5.1, 95% CI 2-sided [-0.9 to 11.0]
Statistical Analysis 2: Comparison: 13vPnC+QIV/Placebo vs Placebo+QIV/13vPnC; Strain A/H3N2: Exact 2-sided CI and corresponding p-value (based on Chan and Zhang) for the difference in proportions, (13vPnC+QIV/placebo - placebo+QIV/13vPnC), expressed as a percentage; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.232, Chan and Zhang method; Percentage Difference = -3.8, 95% CI 2-sided [-9.9 to 2.4]
Statistical Analysis 3: Comparison: 13vPnC+QIV/Placebo vs Placebo+QIV/13vPnC; Strain B/Brisbane: Exact 2-sided CI and corresponding p-value (based on Chan and Zhang) for the difference in proportions, (13vPnC+QIV/placebo - placebo+QIV/13vPnC), expressed as a percentage; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.734, Chan and Zhang method; Percentage Difference = -1.0, 95% CI 2-sided [-6.6 to 4.5]
Statistical Analysis 4: Comparison: 13vPnC+QIV/Placebo vs Placebo+QIV/13vPnC; Strain B/Massachusetts: Exact 2-sided CI and corresponding p-value (based on Chan and Zhang) for the difference in proportions, (13vPnC+QIV/placebo - placebo+QIV/13vPnC), expressed as a percentage; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.627, Chan and Zhang method; Percentage Difference = -1.5, 95% CI 2-sided [-7.2 to 4.3]

11. Secondary Outcome: Geometric Mean Fold Rise (GMFR) in Hemagglutination Inhibition Assay (HAI) 1 Month After Vaccination 1 to Immediately Before Vaccination 1
Description: Fold rise 1 month after Vaccination 1 to before Vaccination 1 was calculated for each influenza virus strain (A/H1N1, A/H3N2, B/Brisbane and B/Massachusetts). GMFRs were calculated using all participants with available data from both the specified blood draws. CI for the GMFRs were back transformations of a CI based on the Student t distribution for mean fold rise. Here, "number of participants analyzed" signifies participants with valid and determinate assay results for specified strain at both the specified blood draws.
Time Frame: Immediately before Vaccination 1, 1 month after Vaccination 1
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: fold rise
Arm/Group | 13vPnC+QIV/Placebo | Placebo+QIV/13vPnC
Number analyzed (Participants) | 427 | 430
fold rise
  Strain: A/H1N1 | 2.4 [2.17 to 2.64] | 2.2 [2.01 to 2.41]
  Strain: A/H3N2 | 2.3 [2.09 to 2.51] | 2.4 [2.15 to 2.59]
  Strain: B/Brisbane | 2.1 [1.97 to 2.32] | 2.2 [1.98 to 2.34]
  Strain: B/Massachusetts | 2.2 [1.98 to 2.34] | 2.1 [1.98 to 2.30]

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as nonserious in another participant, or one participant may have experienced both a serious and nonserious event during the study.
Groups:
- 13vPnC+QIV/Placebo: After Vaccination 1: All participants received 0.5 mL single dose of 13vPnC vaccine intramuscularly along with a dose of QIV (as per official recommendations) intramuscularly at Day 1 (Vaccination 1) followed by 0.5 mL placebo matched to 13vPnC vaccine intramuscularly 1 month after Vaccination 1, were assessed from Vaccination 1 up to before Vaccination 2.
- Placebo+QIV/13vPnC: After Vaccination 1: All participants received 0.5 mL placebo matched to 13vPnC vaccine intramuscularly along with a dose of QIV intramuscular injection (as per official recommendations) at Day 1 (Vaccination 1) followed by 0.5 mL single dose of 13vPnC vaccine intramuscularly 1 month after Vaccination 1, were accessed from Vaccination 1 up to before Vaccination 2.
- 13vPnC+QIV/Placebo: After Vaccination 2: All participants received 0.5 mL single dose of 13vPnC vaccine intramuscularly along with a dose of QIV (as per official recommendations) intramuscularly at Day 1 (Vaccination 1) followed by 0.5 mL placebo matched to 13vPnC vaccine intramuscularly 1 month after Vaccination 1, were assessed from after Vaccination 2 up to before 1 month blood draw after Vaccination 2.
- Placebo+QIV/13vPnC: After Vaccination 2: All participants received 0.5 mL placebo matched to 13vPnC vaccine intramuscularly along with a dose of QIV intramuscular injection (as per official recommendations) at Day 1 (Vaccination 1) followed by 0.5 mL single dose of 13vPnC vaccine intramuscularly 1 month after Vaccination 1, were assessed from after Vaccination 2 up to before 1 month blood draw after Vaccination 2.
- 13vPnC+QIV/Placebo: After 13vPnC Vaccination: All participants received 0.5 mL single dose of 13vPnC vaccine intramuscularly along with a dose of QIV (as per official recommendations) intramuscularly at Day 1 (Vaccination 1) followed by 0.5 mL placebo matched to 13vPnC vaccine intramuscularly 1 month after Vaccination 1, were assessed after 13vPnC Vaccination.
- Placebo+QIV/13vPnC: After 13vPnC Vaccination: All participants received 0.5 mL placebo matched to 13vPnC vaccine intramuscularly along with a dose of QIV intramuscular injection (as per official recommendations) at Day 1 (Vaccination 1) followed by 0.5 mL single dose of 13vPnC vaccine intramuscularly 1 month after Vaccination 1, were assessed after 13vPnC Vaccination.
- 13vPnC+QIV/Placebo: at 6-Month Follow-up: All participants received 0.5 mL single dose of 13vPnC vaccine intramuscularly along with a dose of QIV (as per official recommendations) intramuscularly at Day 1 (Vaccination 1) followed by 0.5 mL placebo matched to 13vPnC vaccine intramuscularly 1 month after Vaccination 1, were assessed from blood draw 1 month blood after Vaccination 2 to 6-month follow-up.
- Placebo+QIV/13vPnC: at 6-Month Follow-up: All participants received 0.5 mL placebo matched to 13vPnC vaccine intramuscularly along with a dose of QIV intramuscular injection (as per official recommendations) at Day 1 (Vaccination 1) followed by 0.5 mL single dose of 13vPnC vaccine intramuscularly 1 month after Vaccination 1, were assessed from blood draw 1 month blood after Vaccination 2 to 6-month follow-up.
Arm/Group | 13vPnC+QIV/Placebo: After Vaccination 1 | Placebo+QIV/13vPnC: After Vaccination 1 | 13vPnC+QIV/Placebo: After Vaccination 2 | Placebo+QIV/13vPnC: After Vaccination 2 | 13vPnC+QIV/Placebo: After 13vPnC Vaccination | Placebo+QIV/13vPnC: After 13vPnC Vaccination | 13vPnC+QIV/Placebo: at 6-Month Follow-up | Placebo+QIV/13vPnC: at 6-Month Follow-up
Serious Adverse Events (participants affected / at risk) | 6/439 | 0/437 | 7/431 | 6/432 | 6/439 | 6/432 | 5/439 | 6/437
Other Adverse Events (participants affected / at risk) | 62/439 | 52/437 | 42/431 | 51/432 | 62/439 | 51/432 | 6/439 | 6/437
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 13vPnC+QIV/Placebo: After Vaccination 1 (N=439) | Placebo+QIV/13vPnC: After Vaccination 1 (N=437) | 13vPnC+QIV/Placebo: After Vaccination 2 (N=431) | Placebo+QIV/13vPnC: After Vaccination 2 (N=432) | 13vPnC+QIV/Placebo: After 13vPnC Vaccination (N=439) | Placebo+QIV/13vPnC: After 13vPnC Vaccination (N=432) | 13vPnC+QIV/Placebo: at 6-Month Follow-up (N=439) | Placebo+QIV/13vPnC: at 6-Month Follow-up (N=437)
Colitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Chest pain (General disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Gangrene (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Localised infection (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Cardiogenic shock (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hiatus hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Osteomyelitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Surgical failure (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bone loss (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 13vPnC+QIV/Placebo: After Vaccination 1 (N=439) | Placebo+QIV/13vPnC: After Vaccination 1 (N=437) | 13vPnC+QIV/Placebo: After Vaccination 2 (N=431) | Placebo+QIV/13vPnC: After Vaccination 2 (N=432) | 13vPnC+QIV/Placebo: After 13vPnC Vaccination (N=439) | Placebo+QIV/13vPnC: After 13vPnC Vaccination (N=432) | 13vPnC+QIV/Placebo: at 6-Month Follow-up (N=439) | Placebo+QIV/13vPnC: at 6-Month Follow-up (N=437)
Angina pectoris (Cardiac disorders) | 0 | 2 | 0 | 1 | 0 | 1 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 2 | 1 | 1 | 2 | 1 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hiatus hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 3 | 3 | 0 | 3 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rectal prolapse (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Injection site pain (General disorders) | 8 | 2 | 0 | 3 | 8 | 3 | 0 | 0
Pyrexia (General disorders) | 0 | 4 | 0 | 1 | 0 | 1 | 0 | 0
Injection site erythema (General disorders) | 2 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Injection site induration (General disorders) | 2 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Injection site swelling (General disorders) | 2 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Vaccination site pain (General disorders) | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Peripheral swelling (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vaccination site reaction (General disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vaccination site induration (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 8 | 4 | 3 | 4 | 8 | 4 | 0 | 0
Bronchitis (Infections and infestations) | 3 | 4 | 4 | 4 | 3 | 4 | 0 | 0
Nasopharyngitis (Infections and infestations) | 3 | 3 | 4 | 1 | 3 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 5 | 1 | 2 | 4 | 5 | 4 | 0 | 0
Sinusitis (Infections and infestations) | 2 | 2 | 1 | 4 | 2 | 4 | 0 | 0
Gastroenteritis (Infections and infestations) | 2 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Tooth abscess (Infections and infestations) | 1 | 1 | 0 | 3 | 1 | 3 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 2 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Abdominal abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 2 | 2 | 0 | 2 | 0 | 0
Fungal infection (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastrointestinal viral infection (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Gingivitis (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Groin infection (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Tooth infection (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Chemical burn of skin (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Chemical burns of eye (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 4 | 2 | 0 | 2 | 1 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 0
Skeletal injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Splinter (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood pressure increased (Investigations) | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 0 | 2 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0 | 1 | 3 | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 3 | 4 | 2 | 0 | 2 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 2 | 0 | 1 | 0 | 0 | 0
Nerve compression (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 1 | 1 | 0 | 1 | 1 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Prostatitis (Reproductive system and breast disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 2 | 0 | 2 | 0 | 0
Haematoma (Vascular disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Atrioventricular block first degree (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vitreous floaters (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Food poisoning (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Loose tooth (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Injection site haematoma (General disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Staphylococcal infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Electrocardiogram T wave abnormal (Investigations) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Lactic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0 | 2 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Balance disorder (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Urine odour abnormal (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Testicular pain (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 0 | 2 | 0 | 0
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cardiomyopathy (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Food allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Chronic sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ovarian cyst (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pelvic haematoma (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Aortic arteriosclerosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 1 | 1 | 0 | 2 | 1 | 2 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.